CLINICAL TRIAL: NCT06350227
Title: Impact of Different Hemostasis Methods on Ovarian Function and Fertility During Laparoscopic Ovarian Cystectomy of Benign Ovarian Cyst
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Yanru Long, Resident physician, West China Second University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WestChinaSU
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Cyst Benign
MeSH Terms: interventions — Sutures; Electrocoagulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- The absorbable hemostat (Experimental)
  Interventions: Combination Product: the absorbable hemostat and suture
- Electrocoagulation (Active Comparator)
  Interventions: Combination Product: electrocoagulation and suture
- Suture alone (Placebo Comparator)
  Interventions: Other: suture

INTERVENTIONS:
Combination Product: the absorbable hemostat and suture — The hemostasis method of the experimental group is to use both the absorbable hemostat and suture.
  Arms: The absorbable hemostat
Combination Product: electrocoagulation and suture — The active comparator group is to use electrocoagulation and suture simultaneously to stop bleeding.
  Arms: Electrocoagulation
Other: suture — The placebo comparator is to use suture alone for hemostasis.
  Arms: Suture alone

SUMMARY:
The purpose of this study is to compare the impact of different hemostasis methods during laparoscopic ovarian cystectomy on ovarian function and fertility in women with benign ovarian cysts.

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed with benign ovarian cysts requiring surgical management.
2. Women who choose laparoscopic ovarian cystectomy voluntarily sign a surgical consent form.
3. Women participating in this study recognize three hemostatic methods and are ready to randomly accept one of them.
4. Women aged between 18 and 40 years old.
5. It was diagnosed by ultrasound as unilateral or bilateral benign ovarian cysts with a maximum diameter of 4-8cm. The nature of the cysts is ultimately confirmed by postoperative pathological examination.
6. Women with no previous history of ovarian surgery, chemotherapy, or pelvic radiation therapy.
7. Patients with no history of endocrine disorders such as hyperprolactinemia, hypothyroidism, or hyperthyroidism, and no history of endocrine therapy within 6 months before laparoscopic ovarian cystectomy.

Exclusion Criteria:

1. Polycystic ovary syndrome.
2. Pregnancy or lactation period.
3. Women with active pelvic inflammatory disease, genital or extragenital malignant tumors.
4. Women who have undergone two or more pelvic or abdominal surgeries.
5. Evidence of premature ovarian failure or premature menopause, such as AMH<1ng/ml.
6. Conversion to open surgery.
7. Women who refuse to sign informed consent or are unable to attend follow-up regularly.
8. Cysts that do not originate from the ovaries or have the characteristics of malignant tumors.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Antral Follicle Count (AFC) | Preoperative quantity and postoperative quantity for 1, 3, and 6 months
  Antral follicle count (AFC) generally refers to the basic follicles in ovaries, which have not yet begun to develop. If the number of AFC is within the normal range (usually 5-10), it indicates that the ovarian reserve function is normal. If the number is low, it generally means that the ovarian reserve function is relatively low. If the number is high, it may be caused by polycystic ovary syndrome. Besides, AFC can be detected through ultrasound examination, and the number of AFC can directly reflect the ovarian reserve of each ovary.

SECONDARY OUTCOMES:
Anti-Mullerian hormone (AMH) | Preoperative level and postoperative level at 1, 3, and 6 months
  Anti-Mullerian hormone (AMH), which can be detected through blood tests, is considered a reliable marker produced by ovarian granulosa cells. The level of AMH indirectly reflects the number of ovarian follicular pools and the joint reserve of both ovaries. In addition, the level of AMH fluctuates less throughout the menstrual cycle. Besides, AMH is almost unrelated to the menstrual cycle and is not affected by gonadotropin-releasing hormone (GnRH) agonists or oral contraceptives.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Sichuan University, Chengdu, Sichuan, China